CLINICAL TRIAL: NCT04767113
Title: A Randomized, Controlled Trial of Continuous Heparin Versus Placebo Infusion to Prevent Catheter-related Thrombosis in Infants After Cardiac Surgery
Brief Title: Continuous Heparin Infusion to Prevent Catheter-related Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GPPH heparin for thrombosis
Record Dates: First submitted 2021-02-06; First posted 2021-02-23 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Surgery; Central Venous Catheter Thrombosis; Heparin
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis | interventions — Heparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Infant participants were blinded naturally, while ultrasonographers for central venous catheter (CVC)-related thrombosis were blinded, especially after interventions were stopped.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin group (Experimental): Continuous infusion of heparin was used to maintain the patency of CVC.
  Interventions: Drug: Heparin sodium
- Control group (Placebo Comparator): Continuous infusion of heparin was used at the corresponding speed.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Heparin sodium — For infants without thrombosis at enrollment, heparin 1 U/kg/h/line for term infants was used and 0.5 U/kg/h/line for preterm infants. The speed of infusion was 0.5ml/h.
  For infants with thrombosis at enrollment, heparin 10-15 U/kg/h for term infants was used with a target activated partial thromboplastin time 60-70s. Other interventions were at the clinical team's discretion under the local protocol.
  Other Names: unfractionated heparin
  Arms: Heparin group
Drug: Normal saline — For infants enrolled, normal saline was infused at the corresponding speed.
  Arms: Control group

SUMMARY:
Catheter-related thrombosis could impair blood flow in the vein, block the central venous catheter, induce catheter-related infection or venous thromboembolism in the deep veins or pulmonary vessels, which furthermore progress into the post-thrombotic syndrome.

Researches using echogenic mass as the primary outcome could miss those premature thrombi which might not be seen on traditional ultrasonography but may be detected by Duplex and Doppler ultrasound with vessel compression. Moreover, studies indicated that some thrombus developed after the catheter removal. Removal of the catheter is not the endpoint of thrombus detection. This study is designed to determine the preventive effects of continuous heparin infusion on real-world central venous catheter-related thrombosis in infants after cardiac surgery.

DETAILED DESCRIPTION:
Catheter-related thrombosis could impair blood flow in the vein, block the central venous catheter, induce catheter-related infection or venous thromboembolism in the deep veins or pulmonary vessels, which furthermore progress into the post-thrombotic syndrome. Researches using echogenic mass as the primary outcome could miss those premature thrombi which might not be seen on traditional ultrasonography but may be detected by Duplex and Doppler ultrasound with vessel compression. Moreover, studies indicated that some thrombus developed after the catheter removal. Removal of the catheter is not the endpoint of thrombus detection. This study is designed to determine the preventive effects of continuous heparin infusion on real-world central venous catheter-related thrombosis in infants after cardiac surgery. One hundred and twenty-four infants were randomized to the intervention group or the control group. Unfractionated heparin or normal saline was infused continuously through each lumen of the central venous catheter at the speed of 0.5 ml/h/line until the catheter was removed. Catheter-related thrombosis was detected by point-of-care Duplex and Doppler ultrasound periodically until 30 days after the cardiac surgery or discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* less than 3 months of age at admission, post-cardiac surgery, with CVC indwelled

Exclusion Criteria:

* parents' refusal, requiring postoperative anticoagulant administration (extracorporeal membrane oxygenation support, prosthetic devices), the contradiction to heparin (coagulopathy or hypercoagulable state, platelet level less than 50000/dL, clinically significant bleeding tendency, allergy to heparin)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
124 infants of CVC-related thrombosis by point-of-care echography or ultrasound | 30 days after cardiac surgery or at discharge, whichever comes first
  CVC-related thrombosis of any catheter as imaged by echocardiogram or ultrasound at 30 days after cardiac surgery. Thrombus was defined as an echogenic mass near the tip of the catheter or slow/no flow detected by Duplex and Doppler ultrasound at the nearby vessels and the on-site vessel couldn't be clasped as narrow as the collateral vessel by compression of the probe.

SECONDARY OUTCOMES:
124 infants of heparin-related comorbidity | 30 days after cardiac surgery or at discharge, whichever comes first
  Abnormal coagulation and hemostasis were defined as treatment initiation by the clinical teams at the discretion of heparin adverse events. Heparin-induced thrombocytopenia was confirmed with consistent low platelet level and positive enzyme-linked immunosorbent assay heparin-platelet factor 4 antibody assay. Catheter-related sepsis was defined as culture of the same organism from both the catheter tip and at least one percutaneous blood culture. Culture of the same organism from the catheter was also accepted as an alternative of culture of catheter tip.

OTHER OUTCOMES:
Post-thrombotic syndrome | 6 months after cardiac surgery
  The symptoms of post-thrombotic syndrome included aching, swelling, itchy and ulcer in the indwelling site and the collateral varicose veins.

CONTACTS AND LOCATIONS:
Overall Officials: Yunxia Sun, MD, Principal Investigator — Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All data published and other related data were available after publication. No private information would be published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the date of publication to 5 years after publication.
Access Criteria: Requests to the corresponding author were necessary.

REFERENCES:
- [Derived] Tan Y, Sun X, Zhong J, Zou Y, Ren Y, Liu Y, Zhao L, Zhuang J, Wang S, Sun Y, Wang Y. A Randomized, Controlled Trial of Continuous Heparin Infusion to Prevent Asymptomatic Catheter-related Thrombosis at Discharge in Infants After Cardiac Surgery: The CHIP-CRT Trial. J Pediatr Hematol Oncol. 2024 Aug 1;46(6):e406-e411. doi: 10.1097/MPH.0000000000002905. Epub 2024 Jun 25. PMID 38934602